CLINICAL TRIAL: NCT01926561
Title: Predicting the Occurence of Hypotensive Bradycardic Events in the Patients Undergoing Arthroscopic Shoulder Surgery in the Sitting Position Under Interscalene Brachial Plexus Block
Brief Title: Predictive Factors for Hypotensive Bradycardic Events During Arthroscopic Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, JongHae Kim, Department of Anesthesiology and Pain Medicine, Daegu Catholic University Medical Center
Other Study IDs: CR-11-072
Record Dates: First submitted 2013-08-14; First posted 2013-08-21 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Syncope, Vasovagal
Keywords: Hypotensive bradycardic event; Interscalene brachial plexus block; Sitting position; Shoulder arthroscopic surgery
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypotensive bradycardic event: The participants are assigned to hypotensive bradycardic event (HBE) group when they experience signs or symptoms associated with syncope, hypotension, or bradycardia, which are treated with vasopressors or inotropics following sitting position after interscalene brachial plexus block is done. Otherwise, they are assigned to non-HBE group.
  Interventions: Other: Interscalene brachial plexus block

INTERVENTIONS:
Other: Interscalene brachial plexus block — After sterile draping around interscalene groove with povidone, a nerve stimulating needle connected to a nerve stimulator is inserted through the interscalene groove. Following involuntary contraction of shoulder, arm, forearm, or hand muscles with 0.5 milliamperes at 1 Hz using the nerve stimulator, 30 to 40 ml of mixture of 1% mepivacaine 20 ml and 0.75% ropivacaine 20 ml are injected.

SUMMARY:
Patients's demographics and perioperative factors affect the occurrence of hypotensive bradycardic events in the patients undergoing arthroscopic shoulder surgery in the sitting position under interscalene block.

DETAILED DESCRIPTION:
Patients' age, Side of the block,Horner's syndrome, the degree of blockade, preoperative fasting time and fluid administration volume, waiting time for sitting position after the block, intraoperative use of opioids and antihypertensives, and change of heart rate variability before the block and after sitting position affect the occurrence of hypotensive bradycardic events in the patients undergoing arthroscopic shoulder surgery in the sitting position under interscalene block.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 80 years
* American Society of Anesthesiologists physical status I-II
* Body mass index < 35 kg/m2

Exclusion Criteria:

* Coagulation deficiencies
* Known allergies to local anesthetics
* Neurologic deficit on the side to be operated
* Inflammation at the puncture site for interscalene brachial plexus block
* Coronary artery disease
* Cardiac conduction disorders and arrhythmias
* Congestive heart disease
* Diabetes mellitus
* Serum electrolyte abnormalities
* Autonomic dysfunction
* Psychiatric disorders
* Patients refusal
* Communications difficulties
* Failure of interscalene brachial plexus block

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are scheduled to receive elective shoulder arthroscopic surgery in the sitting position under interscalene brachial plexus block
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Patient's age and gender, fasting time, administered volume, blood pressure, and heart rate variability | Prior to ISBPB
  Patients'age and gender, preoperative fasting time and volume of fluid administered, pre-block mean arterial pressure and heart rate, logarithmically transformed low frequency, high frequency, and total power of heart rate variability

SECONDARY OUTCOMES:
Side of the block, volume of local anesthetics used, number of patients having Horner's syndrome, hoarseness, and subjective dyspnea, degree of dermatomal and motor blockade | 20 minutes after the end of local anethetics injection
  Side of the block, volume of local anesthetics used, number of patients having Horner's syndrome (ptosis, miosis, and anhidrosis), hoarseness, and subjective dyspnea, degree of dermatomal blockade (C5, C6, C7, C8, and T1), and degree of motor blockade (median, ulnar, radial, and musculocutaneous nerve)
Waiting time for sitting position, heart rate variability, mean arterial pressure, heart rate, frequency of antihypertensives and opioids use, and onset of hypotensive bradycardic events | after the sitting position (expected average of 2 hours including surgery readiness time and duration of surgery)
  Waiting time for sitting position (time from the end of interscalene brachial plexus block to the sitting position), logarithmically transformed high frequency, low frequency, and total power of heart rate variability, mean arterial pressure, heart rate, frequency of intraoperative use of antihypertensives and opioids, and onset of hypotensive bradycardic events

CONTACTS AND LOCATIONS:
Overall Officials: WoonSeok Roh, Doctor, Study Chair — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

REFERENCES:
- [Background] Simeoforidou M, Vretzakis G, Chantzi E, Bareka M, Tsiaka K, Iatrou C, Karachalios T. Effect of interscalene brachial plexus block on heart rate variability. Korean J Anesthesiol. 2013 May;64(5):432-8. doi: 10.4097/kjae.2013.64.5.432. Epub 2013 May 24. PMID 23741566
- [Background] Song SY, Roh WS. Hypotensive bradycardic events during shoulder arthroscopic surgery under interscalene brachial plexus blocks. Korean J Anesthesiol. 2012 Mar;62(3):209-19. doi: 10.4097/kjae.2012.62.3.209. Epub 2012 Mar 21. PMID 22474545
- [Background] Sia S, Sarro F, Lepri A, Bartoli M. The effect of exogenous epinephrine on the incidence of hypotensive/bradycardic events during shoulder surgery in the sitting position during interscalene block. Anesth Analg. 2003 Aug;97(2):583-588. doi: 10.1213/01.ANE.0000070232.06352.48. PMID 12873958
- [Background] Liguori GA, Kahn RL, Gordon J, Gordon MA, Urban MK. The use of metoprolol and glycopyrrolate to prevent hypotensive/bradycardic events during shoulder arthroscopy in the sitting position under interscalene block. Anesth Analg. 1998 Dec;87(6):1320-5. doi: 10.1097/00000539-199812000-00020. PMID 9842820